CLINICAL TRIAL: NCT01030146
Title: Management of Allergic Rhinitis Patients With Nasal Steroids and NeilMed® Sinus Rinse™ System With Isotonic Saline: A Prospective Pilot Study
Brief Title: Management of Allergic Rhinitis Patients With Nasal Steroids and NeilMed® Sinus Rinse™ System With Isotonic Saline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: NeilMed Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sinus Rinse
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2014-08

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeilMed® Sinus Rinse™ System (Other): NeilMed® Sinus Rinse™ System with Isotonic Saline twice a day
  Interventions: Drug: NeilMed® Sinus Rinse™ System with Isotonic Saline

INTERVENTIONS:
Drug: NeilMed® Sinus Rinse™ System with Isotonic Saline — NeilMed® Sinus Rinse™ System with Isotonic Saline twice a day

SUMMARY:
You are being asked to volunteer for a research study. You are being asked to participate in this study because you have completed at least one month of drug treatment with a nasal steroid and allergy testing and still have symptoms. This research study is sponsored by NeilMed Pharmaceuticals, Inc. The purpose of this study is to compare quality of life outcomes in patients who continue medical treatment plus the use of the NeilMed Sinus Rinse low-pressure pump with saline. Your participation in this study may help to improve the management of patients with allergic rhinitis.

Allergic rhinitis is a common health problem, affecting between 10% and 40% of the world's population. Presently, antihistamines and nasal steroids are the standard treatment for allergic rhinitis. To further clarify these findings, we propose a study comparing the differences in quality of life improvements, by using a series of questionnaires, between subjects electing continued medical management and those electing medical treatment plus nasal wash.

The investigators in charge of the study are Dr. Rodney J. Schlosser and Dr. Shaun A. Nguyen. Approximately 40 patients will be enrolled in this study at the Medical University of South Carolina (MUSC Hospital). You will have the choice of choosing either to receive only medical treatment or to receive medical treatment with nasal wash.

DETAILED DESCRIPTION:
Before you are allowed to participate in this study, the doctor will review your medical history and ask you questions to see if you qualify for the study.

This study follows the standard of care in managing patients with allergic rhinitis. You will undergo allergy testing with the skin prick test (SPT), a baseline NPIF (Nasal Peak Inspiratory Flow, where we ask you to breath in a mask) measurement, and a baseline assessment with the mRQLQ (Mini Rhinoconjunctivitis Quality of Life Questionnaire) questionnaire. You will be asked to continue drug treatment with nasal steroid along with the NeilMed Sinus Rinse low-pressure pump with isotonic saline as an add-on treatment. You will be given supplies and instructions on the use of the NeilMed Sinus Rinse low-pressure pump with saline to be performed twice a day for two months. You will be asked to come back at the end of 1 month and 2 months, where you will complete another mRQLQ and NPIF assessment. In addition, you will be asked to return low-pressure nasal irrigation bottle for testing of bacteria and fungi at the end of 1 month and 2 months. This is a safety assessment for back wash contamination.

If you are unable to return for scheduled clinic visits, questionnaires will be mailed with self-addressed stamped envelopes with follow-up phone calls to ensure study compliance and minimal attrition C. Duration The time to answer the survey questionnaires will take no longer than 20 minutes on each visit. The entire duration of the study is no longer than 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* male or female adults (aged 18-99) diagnosed with rhinitis who have completed one month of pharmacotherapy exclusively with nasal steroids and allergy testing.

Exclusion Criteria:

* male and female adults who have been diagnosed with sinusitis, cystic fibrosis, or immune deficiency or those unable or unwilling to perform saline irrigations for two months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
mRQLQ | 8 weeks

SECONDARY OUTCOMES:
Nasal Peak Inspiratory Flow | 8 weeks
Safety and Adverse Effects | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rodney J Schlosser, MD, Principal Investigator — Medical University of South Carolina; Shaun A Nguyen, M.D.,CPI, Principal Investigator — Medical University of South Carolina
Locations (1):
- Sinus Center - Medical Univesity of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Nguyen SA, Camilon MP, Schlosser RJ. Identification of microbial contaminants in sinus rinse squeeze bottles used by allergic rhinitis patients. World J Otorhinolaryngol Head Neck Surg. 2019 Jan 5;5(1):26-29. doi: 10.1016/j.wjorl.2018.12.001. eCollection 2019 Mar. PMID 30775698
- [Derived] Nguyen SA, Psaltis AJ, Schlosser RJ. Isotonic saline nasal irrigation is an effective adjunctive therapy to intranasal corticosteroid spray in allergic rhinitis. Am J Rhinol Allergy. 2014 Jul-Aug;28(4):308-11. doi: 10.2500/ajra.2014.28.4066. Epub 2014 May 22. PMID 24857280
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pubmed/24857280